CLINICAL TRIAL: NCT02497573
Title: Study of Diffusion Weighted MRI as a Predictive Biomarker of Response During Radiotherapy for High and Intermediate Risk Squamous Cell Cancer of the Oropharynx (MeRInO Study)
Brief Title: Can DW MRI Predict Outcome During Radiotherapy for Head and Neck Cancer?
Acronym: MeRInO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN15ON249
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Diffuse Weighted MRI — The DW MRI scans will be used to measure ADC and to calculate change in ADC between the 2 scans. Each scan will take approximately 30 minutes. Images will be acquired and analysed as per the separate scanning protocol.

SUMMARY:
Around 50% of patients with locally advanced H&N cancer fail to achieve loco-regional control. Currently it cannot be predicted, during treatment, who will fall into this group of non-responders.

This study is designed to assess the value of DW MRI as a predictive biomarker of response to radiotherapy in intermediate and high risk OPSCC.

DETAILED DESCRIPTION:
Around 1000 patients with new cancers of the head and neck (H&N) are registered in Scotland annually. Approximately 60% of these are managed in the west of Scotland. Unfortunately a large proportion, around 60%, of H&N cancers present with locally advanced but non-metastatic disease. These are associated with poor outcomes with 3 year survival around 50%. Despite intensive radical therapy associated with significant acute toxicity, there is a high recurrence rate (up to 50%) and unlike many other cancers, the vast majority of these recurrences, around 80%, occur locally and many patients go on to die from their local disease without developing distant metastases. Locally recurrent tumours cause significant morbidity and palliation is difficult. There is a therefore a clear need to further improve local disease control, both to increase cure rates and to improve quality of life.

This study is designed to assess the value of DW MRI as a predictive biomarker in intermediate and high risk OPSCC. DW MRI and changes in ADC have been shown to correlate with response to treatment in prospective and retrospective studies in SCC H&N. These studies have included all H&N sub-sites with no differentiation between biological sub-types. This study may therefore validate the use of DW MRI as a predictive biomarker specifically in the intermediate and high risk groups of OPSCC. If change in ADC during RT is found to be predictive of eventual clinical outcome and a discriminatory threshold rise in ADC identified, this information could be used to inform treatment intensification in patients responding poorly to RT. This would form the basis of subsequent clinical trials.

The hypothesis of this study is that quantitative DW MRI - i.e. change in ADC during RT - is predictive of locoregional control in intermediate and high risk OPSCC and that a threshold can be identified in ADC change that will discriminate responders from non-responders to radiotherapy.

The design is a single centre observational study to assess the value of DW MRI as a predictive biomarker in HPV-OPSCC. 2 DW MRI scans will be carried out on participants in addition to all standard imaging and procedures for radiotherapy. The information gained from the MRI scans will not be used to change standard treatment for these patients. DW MRI_1 will be obtained prior to radiotherapy commencing. DW MRI_2 will be carried out during the third week of radiotherapy treatment. The DW MRI scans will be used to measure ADC and to calculate change in ADC between the 2 scans. The MRI scans will be carried out during routine hospital visits for radiotherapy planning and treatment therefore will involve no extra visits for participants.

After completion of (chemo) radiotherapy, patients will attend the Beatson WoSCC for follow up visits as per standard protocol at 3, 6, 12, 18 months post treatment. Information regarding recurrence will be collected at these routine visits. No extra post-treatment visits are therefore required from participants.

The recruitment phase is estimated to last for 2 years and patients will be followed up will be for 18 months after completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HPV negative SCC oropharynx or patients with HPV positive SCC oropharynx and a significant smoking history
* Stage III or Iva or IVb disease
* Scheduled to undergo radical radiotherapy or chemo radiotherapy as primary treatment
* 18 years of age or older
* Able to give written informed consent
* Patients willing and able to comply with the protocol for the duration of the study

HPV status: As defined by the Scottish HPV reference laboratory, multiplex assay on Luminex technology Significant smoking history definition: greater than 10 pack years

Exclusion Criteria:

* Head and neck cancers from sub sites other than oropharynx
* HPV+OPSCC in patients with no significant smoking history (low risk OPSCC)
* Patients receiving cetuximab-radiotherapy
* Confirmed distal metastatic disease (stage IVc)
* Patients who have undergone primary surgery for SCC H&N, neck dissection alone permitted
* Patients who have received induction chemotherapy prior to definitive treatment
* Patients with contra-indications to MRI scanning

Contra-indications to MRI:

As per standard diagnostic imaging protocol - cardiac pacemaker, surgery within 8 weeks, aneurysm clipped/treated, metal fragments in eye, previous cranial surgery, any metal in the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate or high risk oropharyngeal squamous cell carcinoma (OPSCC), scheduled to undergo either radiotherapy or chemoradiotherapy as primary treatment in the Beatson West of Scotland Cancer Centre may be suitable for study participation. Suitable patients will be identified at MDT meetings or from the radiotherapy bookings database and approached by the direct clinical care team as they attend for radiotherapy planning appointments. 80 patients will be recruited to the study.
  Each patient will have at least one target lesion (either lymph node or primary site) for ADC analysis and clinical follow up. MnayMany patients will have 2 or more target lesions. The total number of target lesions is therefore highly likely to be greater than 80.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
change in composite ADC | 3 weeks
  Apparent Diffusion Coefficient measured at each MRI for each target lesion and the % change in each target lesion will be recorded at MRI2, in comparison with MRI1
Relapse status | 18 months
  Relapse status (control or failure), for each target lesion, will be recorded at the 18 month time point and compared with baseline. Control is defined as absence of any new mass, serial reduction in size or unchanged size of residual mass. Failure is defined as biopsy proven recurrence, new mass or serial increase in size of residual mass.

SECONDARY OUTCOMES:
Time to Relapse | Up to 22 Months
  If relapse occurs (failure), the time to relapse, from baseline, will be recorded. Failure is defined as biopsy proven recurrence, new mass or serial increase in size of residual mass.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Paterson, PhD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No